CLINICAL TRIAL: NCT01855672
Title: A Multicenter, Randomized, Controlled, Double-Blind, Proof-of-Concept Study Assessing the Safety and Effectiveness of a Signal Generator Device (NMS EBox) for the Treatment of Chronic Migraine
Brief Title: Occipital Nerve Stimulation in the Treatment of Migraine
Acronym: Verona
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business strategic decision not related to safety.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESC-13-001
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-06

CONDITIONS: Migraine
Keywords: Migraine, occipital nerve, stimulation
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perceivable Stimulation (Active Comparator): Stimulation of the occipital nerves.
  Interventions: Device: Stimulation of the Occipital Nerves
- Non-Perceivable (Active Comparator): Stimulation of the occipital nerves.
  Interventions: Device: Stimulation of the Occipital Nerves

INTERVENTIONS:
Device: Stimulation of the Occipital Nerves — Electrical stimulation of the occipital nerves.

SUMMARY:
The objective of this proof-of-concept study is to generate initial safety and effectiveness data for the neuro-modulation stimulation (NMS) E-Box in patients with chronic migraine in an acute setting. The results of this study will determine if further development of this device in a larger study is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 and ≤ 65 years of age females or males;
2. Willing to participate in the study and to complete all study-related procedures, evaluations, and headache diaries;
3. Able to understand, agree to, and sign the study's IRB-approved informed consent form;
4. Has a physician-made diagnosis of Chronic Migraine as defined by the following (a, b, and c):

   1. Headache (tension-type and/or migraine) lasting a minimum of 4 hours on ≥15 days per month for at least 3 months and on ≥XX (redacted by sponsor to preserve integrity of study) days in the 30 days prior to the Screening Visit;
   2. Headaches on ≥8 days per month for at least 3 months that have fulfilled the following:

   i. Headaches with at least two of the following:
   * unilateral location;
   * pulsating quality;
   * moderate or severe pain intensity;
   * aggravation by or causing avoidance of routine physical activity (e.g. walking or climbing stairs);

   ii. AND at least one of the following:
   * nausea and/or vomiting;
   * photophobia and phonophobia;

   iii. OR headaches that have been treated and relieved by triptan(s) or ergot before the expected development of the symptoms listed in 4.b.i and 4.b.ii above;

   c. Headaches are not attributed to a substance or substance withdrawal, infection, cranial neuralgias, cluster headaches, autonomic cephalalgias, or cranial, cervical vascular, non-vascular, intracranial homeostasis and psychiatric disorders;
5. If taking medication (prescribed or over-the-counter) for migraine prophylaxis, the medication must have been taken for at least 2 months and the dosage(s) must have been stable for at least 1 month prior to the Screening Visit. There must be no plan to add to, discontinue, or change the dose of these medications throughout the subject's participation in the study;
6. To be eligible for the inpatient Treatment Period: the subject must have recorded in the Headache Diary ≥XX (redacted by sponsor to preserve integrity of study) headaches days (at least 4 hours of continuous head pain per headache day) in the 30 days immediately prior to the Inpatient Treatment Eligibility Visit (Visit 2);
7. To be eligible for the inpatient Treatment Period: mean head pain severity of ≥XX (redacted by sponsor to preserve integrity of study) and ≤XX (redacted by sponsor to preserve integrity of study) based on the 11-point Numerical Rating Scale (NRS) in the 30 days immediately prior to the Inpatient Treatment Eligibility Visit (Visit 2) [only data from headache days will be used to calculate the mean head pain severity; missing data on a headache day will be considered to be zero (0) for this calculation]; and
8. To be eligible for the inpatient Treatment Period: The subject must be experiencing head pain on the day of the inpatient Treatment Eligibility Visit (Visit 2). Subjects may continue the Screening Period for another week if head pain is not present at Visit 2.

Exclusion Criteria:

1. Any head pain, including coexisting head pain, not attributable to Chronic Migraine as defined in this study's Inclusion Criterion #4;
2. Any condition that could affect the subject's ability to assess the effect of neurostimulation or in which neurostimulation may be a safety concern, including but not limited to:

   1. Known history of epilepsy or recurrent seizures;
   2. Known neurogenic and neuromuscular disorders (i.e. myasthenia gravis, multiple sclerosis, autonomic disorders);
   3. Uncontrolled diabetes mellitus;
   4. Known peripheral neuropathy;
3. History of taking the following medications in the 30 days prior to the Screening Visit:

   1. Opioid and opioid-containing medications;
   2. Butalbital, butalbital-containing, and barbiturate medications;
   3. Systemic corticosteroids (exceptions: acute corticosteroid medication including inhaled therapy (pulmonary), ocular therapy, or non-spinal intra-articular therapy);
4. Urine drug screen that is positive for any of the tested drugs (i.e., cannabis, opiates, barbiturates, amphetamines , benzodiazepines and cocaine) at the Screening Visit (Visit 1) and the Inpatient Treatment Eligibility Visit (Visit 2);
5. Positive pregnancy test at the Screening Visit (Visit 1) or at the Inpatient Treatment Eligibility Visit (Visit 2);
6. Known history of cardiac conduction or heart rate abnormalities associated with symptoms;
7. Uncontrolled hypertension;
8. Any tattoos or extensive tissue scarring in the cervical/occipital area;
9. Any active skin lesions, skin damage, broken skin, history of easy bruising or bleeding disorders, or history of surgery and/or trauma in the cervical/occipital area at the time of the Screening Visit;
10. History of occipital nerve (ON) block, peripheral ON stimulation, or botulinum toxin (e.g., Botox) for treatment of headaches within the 90 days prior to the Screening Visit;
11. Radiofrequency rhizolysis involving the occipital nerve or cervical nerves;
12. Surgery involving the occipital nerve or cervical nerves (e.g. neurectomy or rhizotomy), or cervical ganglionectomy;
13. History of craniotomy or intracranial surgery;
14. Presence of metallic implant (e.g., metal pin, staple, clip) in the skull or neck area;
15. Presence of any implanted neuromodulation or cardiac device;
16. Severe or uncontrolled psychiatric disorders (i.e. schizophrenia, depression, anxiety, or at investigator discretion);
17. Any other medical condition, concomitant medication or finding for which, at the discretion of the investigator, the subject should be excluded for reasons of safety or capacity for study compliance; or
18. Participation in any other clinical study (not to include registries or survey-only studies) within 30 days or 5 half lives of an investigational drug, whichever is longer, of Visit 1 (Screening Visit) and for the duration of the study.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Reduction of Head Pain Severity | Over 96-hours treatment period
  The primary endpoint is overall reduction of head pain severity in subjects with chronic migraine who are treated with the NMS E-Box over a 96-hour treatment period.

SECONDARY OUTCOMES:
Rates of Reduction in Severity of Head Pain | Over the 96-hour treatment period
  Responder rates for reduction in the severity of head pain associated with chronic migraine over the 96-hour Treatment Period (e.g., 30% and 50% responder rates).
Time with No Head Pain | Over the 96-hour Treatment Period
  Increase in cumulative time with no head pain over the 96-hour Treatment Period.
Presence of Symptoms | Over the 96-hour treatment period
  Decrease in the presence of each of the following migraine-associated symptoms (i.e., nausea or vomiting; photophobia; phonophobia) over the 96-hour Treatment Period.
Severity of Symptoms | Over the 96-hour treatment period
  Decrease in the severity of each of the following migraine-associated symptoms (i.e., nausea or vomiting; photophobia; phonophobia) over the 96-hour Treatment Period.
Use of Medication | Over the 96-hour treatment period
  Decrease in the use of any over-the-counter or prescription medication taken for the acute treatment of migraine or head pain over the 96-hour Treatment Period.
Impairment | Over the 96-hour treatment period
  Decrease in Migraine-Related Impairment over the 96-hour Treatment Period.
Sleep Quality | Over the 96-hour treatment period
  Improvement in Sleep Quality over the 96-hour Treatment Period.
PGIC | End of the 96-hour treatment period
  Improvement in the Patient Global Impression of Change (PGIC) for Chronic Migraine at the end of the 96-hour Treatment Period.
CGIC | End of the 96-hour treatment period
  Improvement in the Clinician Global Impression of Change (CGIC) for Chronic Migraine at the end of the 96-hour Treatment Period.
PGIC Migraine | End of the 96-hour treatment period
  Improvement in the Patient Global Impression of Change for Migraine-Related Impairment at the end of the 96-hour Treatment Period.
PGIC Sleep | End of the 96-hour treatment period
  Improvement in the Patient Global Impression Change for Sleep Quality at the end of the 96-hour Treatment Period.

OTHER OUTCOMES:
Safety | Over the treatment and follow-up periods
  The safety endpoint is to further characterize the safety profile of the NMS E-Box through the collection and evaluation of adverse events. The occurrence of adverse events will be compared between arms.

CONTACTS AND LOCATIONS:
Overall Officials: David Biondi, DO, Study Director — Janssen, LP; Jeff Hammond, MD, Study Director — Ethicon, Inc.
Locations (4):
- United States (4):
  - ActivMed, Newington, New Hampshire
  - Clinilabs, New York, New York
  - Community Research, Cincinnati, Ohio
  - TJU, Philadelphia, Pennsylvania